CLINICAL TRIAL: NCT02770339
Title: Pharmacogenomic Profiling of Pediatric Patients on Psychotropic Medications in an Emergency Department
Brief Title: Pharmacogenomic Profiling of Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pallavi Ghosh, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F160225002
Record Dates: First submitted 2016-05-07; First posted 2016-05-12 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Mental Disorders; Metabolism Medication Toxicity; Pediatric Disorder
Keywords: Pharmacogenomics; Psychiatric crisis; Drug overdose; Psychotropic medications
MeSH Terms: conditions — Mental Disorders; Drug Overdose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to store DNA for potential Genomic Data Sharing (GDS)( studies if further study is prompted by the results of this study.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the proportion of children presenting to a pediatric emergency department with an acute mental health/behavioral crisis or clinical drug toxicity who have a "match" or "mismatch" between the genes for drug metabolizing enzymes and their current or recent drug therapy. The investigators will utilize a readily available and FDA-approved cheek swab DNA test --GeneSight®--in these children that categorizes patients into 3 different type of groups - RED, YELLOW, and GREEN based on individuals' abilities to metabolize psychotropic drugs . Specific objectives include:

* The relationship of genomic mismatch to serum drug concentrations, either low or high
* The proportion of children with a genomic mismatch who present to PED with intentional self-injury.
* The relationship between match versus mismatch and self- and caregiver-reported outcomes of functioning, drug efficacy, and drug tolerability.
* Examine the proportion of children/adolescents who present to PED with an adverse drug reaction to one or more psychotropic with a genomic mismatch.
* Quantify the specific adverse reactions related to a mismatch of genotypes.

DETAILED DESCRIPTION:
Background:

The Centers for Disease Control and Prevention estimate that 13-20% of children living in the United States experience a mental disorder in a given year and an estimated $247 billion is spent each year on childhood mental disorders. In the last 5 years, emergency departments (ED) have been facing dramatic increases in the volume of pediatric patients presenting for evaluation and treatment of mental and behavioral disorders, to the point where it has been termed a national pediatric mental health crisis. Coincident with this increase has been the exponential increase in the number of children, both children as young as 2 years of age and adolescents, being prescribed 1 or more psychotropic medications-antidepressants (AD), antipsychotics (AP), and medications for Attention Deficit Hyperactivity Disorder (ADHD)-- for various mental and behavioral disorders in the last 10 years. More intentional overdoses, therapeutic errors, and/or adverse drug reactions (ADR) to these classes of medications are being evaluated in our pediatric emergency department (PED), potentially attributable to the increased number of children taking these medications. National Poison Data System (NPDS) -reported exposures to these medication classes continue to increase in both children and adolescents.

Numbers and rates of adverse drug event (ADE) emergency department visits involving psychiatric medications among US adults are significant, although the numbers in children are less well defined. The development of adverse medical conditions related to antipsychotic and other psychotropic medication use in children and adolescents has been found to be significantly associated with higher total costs of health care and to higher utilization of outpatient, emergency, and inpatient services over time.

Interindividual differences of people's clinical responses to psychotropic drugs and adverse drug reactions despite identical disease severity or etiology may be better explained by genetic variation among patients than other various factors. We will determine if genetic polymorphisms for genes coding for CYP450 drug metabolizing enzymes are associated with therapeutic failures and/or toxicity using the GeneSight® buccal swab test. Multiple published adult clinical studies have demonstrated that this combinatorial, multi-gene test better predicts antidepressant treatment outcomes for patients with depression and their use of health care resources, than any of the individual genes that comprise the test. One study demonstrated 70% greater improvement in depressive symptoms when GeneSight® guided physicians' treatment compared to unguided treatment, while another demonstrated a 67% increase in total healthcare visits when medication plans did not match their genetic profiles, contributing to significant increase in healthcare costs.19,20 Recent recommendations from the Clinical Pharmacogenetics Implementation Consortium of the National Institutes of Health Pharmacogenomics Research Network suggest that current data indicate that genotypes for CYP2D6 and CYP2C19 can lead to specific treatment recommendations.

To the investigators knowledge, this study is one of the first to propose the use of pharmacogenomic tests to study toxicity or treatment failure in pediatric patients using psychotropic medications and assess its clinical utility in patients presenting in crises to an ED. The results of this study are very likely to change clinical practice leading to increased pharmacogenomic testing of children and adolescents at their point of care in outpatient clinics, inpatient services, or PEDs. If successful, this project will lay the groundwork for future prospective analyses of genotypic "match" versus "mismatch" and either symptomatic or toxic adverse outcomes in this cohort presenting to a PED compared to a control population in an outpatient setting.

Study population: Inclusion criteria: Two categories of PED patients on psychotropic medications will be included in this trial: (1) Children/adolescents who present with psychiatric/behavioral crisis or intentional overdose. This would include those referred for psychiatric evaluation, who may have behavioral problems (aggressive behavior, violent behavior), suicidal or homicidal thoughts, recent history of self-injury (with or without suicidal intent), depression, psychosis, anxiety, altered mental status, or violence. 2) Children/adolescents who present to the PED with a suspected adverse drug reaction to any of the psychotropic/ADHD medications (toxicity)

Exclusion criteria: (1) Patients on the aforementioned medications who present to the PED with a chief complaint other than those listed above. (2) Participants who present with acute intoxication with alcohol or drugs of abuse. (3) Patients in Alabama Department of Human Resources (DHR) custody. (4) Those with medical conditions that preclude participation. (5) Those with previous pharmacogenomic testing.

Methods:

The investigators will enroll 100 patients 3-18 years of age who are taking 1 or more AD, AP, and/or ADHD medication presenting to the PED at Children's of Alabama with mental health/behavioral crisis and/or adverse drug reaction to one of these drugs. This would include those referred for psychiatric evaluation, who may have behavioral problems, suicidal or homicidal thoughts, recent history of self-injury (with or without suicidal intent), depression, psychosis, anxiety, altered mental status, or violence.

The informed consent process will take place before any study-specific procedures are initiated. Signed and dated written informed consent must be obtained from each patient/parent/legal caregiver prior to enrollment into the study. Assent for patients 7-13 years of age will be obtained unless criteria for waiver is met.

Data Collection

Buccal Swab: GeneSight uses a combinatorial psychiatric pharmacogenomics (CPGx) multi-gene approach to produce a personalized interpretive report that categorizes psychotropic medications into three groups (RED [use with increased caution and with more frequent monitoring], YELLOW[use with caution], GREEN[use as directed) based on objective, evidence-based gene-drug interactions. This decision support tool helps clinicians to make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications. It consists of a cotton swab. GeneSight Psychotropic provides information on 38 FDA-approved antidepressant and antipsychotic drugs. GeneSight® ADHD provides information on 100% of the FDA-approved medications for ADHD.

Blood Sampling: Blood for measuring serum concentrations of the medications that the patient is taking will be obtained (15-20 ml depending on how many medications the child is taking, 10 ml if the patient is < 14 kg). A small portion of this blood (5 ml) will also be banked for future DNA genomic analyses. These blood volumes are all within accepted volumes for patients in this age range.

Note: Blood samples are normally obtained in patients with drug overdose, suspected drug toxicity as part of their standard evaluation as well as many patients being admitted to an inpatient psychiatric facility.

12-lead Electrocardiogram: Rate, rhythm, QRS interval, QT, corrected QT interval (QTc), terminal R wave in lead aVR will be recorded. The ECG is usually a standard part of the evaluation for ingestions/overdose/suspected drug toxicity and sometimes for patients being admitted to an inpatient psychiatric facility.

In addition to these tests we will also collect: (1) Demographics: age, sex/gender, race/ethnicity, living situation, educational attainment. (2) Medication History: list of current and past psychotropic medication treatments including name, doses, start and stop dates, and estimated response. (3) All other medications. (4) Socioeconomic information, including third party reimbursement. (5) Recall of healthcare utilization over the previous 12 months including hospitalization or ED visits. (6) Indication for psychotropic medication (note that formal diagnostic interviewing will not be performed because of constraints of the ED setting). (7) Reason for the current ED visit (e.g., anxiety, panic attack, intentional self-injury including suicide attempt, suicidal ideation, homicidal ideation, medication overdose, harm to persons or property, other aggression, psychosis, severe depression, other psychiatric cause, adverse drug reaction). (8) Global Assessment of Function (GAF) scale, Clinical Global Impression Scale (CGI-I), and Clinical Global Efficacy Index (CGI-E), all validated scales used extensively in psychiatric research and (9) Clinical toxicity/adverse drug reactions.

Note that the scales delineated in #8 ask for information that is usually part of the physician's history and patient assessment: - self-assessment or the parent/caregiver's assessment of the patient's overall functioning, drug tolerability, drug efficacy. This information has been developed into validated scales.

The process is designed to be relatively brief to allow the study to proceed within the workflow of the PED. Some information will be obtained from the electronic medical record (drug names, duration of therapy, previous psychiatric diagnoses) if the patient, parent, and/or caregiver is unsure or doesn't know.

Statistical Analyses:

* Descriptive statistics, specifically proportions, will be calculated for: Mismatch of proportion of children presenting to PED with GeneSight RED or YELLOW categories and i.) acute psychiatric/behavioral crisis ED visits; ii.) serum drug concentrations, high or low; and iii.) overdose of drugs.
* Frequency of self-reported/caregiver-reported negative scores on GAF (score 5,6,7), CGI-I (score 5,6,7), CGI-E scores
* Relationship between Mismatch(RED,YELLOW) and Match (GREEN) and self- and/or care-reported GAF, CGI-I, CGI-E scores
* Descriptive statistics, specifically proportions will be calculated for: Mismatch of proportion of children presenting to PED with GeneSight genotype RED or YELLOW categories and adverse drug reactions
* Frequency of GeneSight genotype mismatch RED or YELLOW categories and specific adverse reactions/clinical toxicity

ELIGIBILITY:
Inclusion Criteria:

* Children taking 1 or more antidepressant, antipsychotic, and/or attention deficit hyperactivity disorder medications.
* Children/adolescents who present with psychiatric/behavioral crisis or intentional overdose. This would include those referred for psychiatric evaluation, who may have behavioral problems (aggressive behavior, violent behavior), suicidal or homicidal thoughts, recent history of self-injury (with or without suicidal intent), depression, psychosis, anxiety, altered mental status, or violence.
* Children/adolescents who present to the PED with a suspected adverse drug reaction to any of the psychotropic/ADHD medications (toxicity).

Exclusion Criteria:

* Patients on the aforementioned medications who present to the PED with a chief complaint other than those listed in the inclusion criteria.
* Participants who present with acute intoxication with alcohol or drugs of abuse.
* Patients in Alabama Department of Human Resources (DHR) custody.
* Those with medical conditions that preclude participation.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects ages 3-18 years of age who present to the pediatric emergency department with an acute psychiatric /behavioral crisis who are also on 1 more psychotropic medications (antidepressants, antipsychotics, attention deficit hyperactivity disorder medications) will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Psychiatric/Behavioral Crisis in Pediatric Emergency Department Genomic Mismatch | Test result will be analyzed within 1 week of patient being enrolled
  The proportion of children presenting with psychiatric/behavioral crises in the PED who have a drug-genotype mismatch
Drug Concentration Genomic Mismatch | Drug concentrations will be measured within 3 months of enrollment
  The relationship between genomic mismatch in drug metabolizing enzymes and abnormal serum drug concentrations (either low or high).
Global Assessment of Functioning/Efficacy of Medications Genomic Mismatch | Analysis of assessment scales/scores with pharmacogenomic test results will occur after enrollment is completed, average of 1 year
  The relationship between negative self- and caregiver-reported outcomes (global assessment of functioning, efficacy of medications) and genotype mismatch.
Overdose of Drugs Genomic Mismatch | Analysis of the association of subjects presenting with drug overdose with pharmacogenomic test results will occur after enrollment is completed, average of 1 year
  The proportion of children/adolescents who present to PED with an overdose and psychotropic drug mismatch.

SECONDARY OUTCOMES:
Adverse Drug Reactions - Therapeutic Dose Genomic Mismatch | Analysis of association between adverse drug reaction and genomic mismatch will occur after enrollment is completed, average of 1 year
  The proportion of children/adolescents who present to PED with adverse drug reaction(s) to one or more who have a genomic mismatch with their psychotropic drugs.
Clinical Toxicity Genomic Mismatch | Analysis of any association between any clinical medication toxicity and genomic testing will occur after enrollment is completed, average of 1 year.
  To quantify the specific adverse reactions related to a mismatch of genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi Ghosh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Based on the initial results with the GeneSight data, the researchers will decide if further analysis (genotype) of the DNA will be undertaken. The informed consent allows the participant to agree or disagree to having their blood stored for this additional analysis. Their decision does not affect their ability to participate in the research study. No personal identifiers will be associated with this analysis. If further analysis is done, the plan is to share through the NIH Genome Data Sharing program, according to its process.

REFERENCES:
- [Background] Pittsenbarger ZE, Mannix R. Trends in pediatric visits to the emergency department for psychiatric illnesses. Acad Emerg Med. 2014 Jan;21(1):25-30. doi: 10.1111/acem.12282. Epub 2013 Dec 6. PMID 24552521
- [Background] Olfson M, King M, Schoenbaum M. Treatment of Young People With Antipsychotic Medications in the United States. JAMA Psychiatry. 2015 Sep;72(9):867-74. doi: 10.1001/jamapsychiatry.2015.0500. PMID 26132724
- [Background] Olfson M. Surveillance of adverse psychiatric medication events. JAMA. 2015 Mar 24-31;313(12):1256-7. doi: 10.1001/jama.2014.15743. No abstract available. PMID 25803347
- [Background] Braga-Neto MB, Warren CA, Oria RB, Monteiro MS, Maciel AA, Brito GA, Lima AA, Guerrant RL. Alanyl-glutamine and glutamine supplementation improves 5-fluorouracil-induced intestinal epithelium damage in vitro. Dig Dis Sci. 2008 Oct;53(10):2687-96. doi: 10.1007/s10620-008-0215-0. Epub 2008 Mar 6. PMID 18320312
- [Background] Altar CA, Carhart JM, Allen JD, Hall-Flavin DK, Dechairo BM, Winner JG. Clinical validity: Combinatorial pharmacogenomics predicts antidepressant responses and healthcare utilizations better than single gene phenotypes. Pharmacogenomics J. 2015 Oct;15(5):443-51. doi: 10.1038/tpj.2014.85. Epub 2015 Feb 17. PMID 25686762
- [Background] Winner JG, Carhart JM, Altar CA, Goldfarb S, Allen JD, Lavezzari G, Parsons KK, Marshak AG, Garavaglia S, Dechairo BM. Combinatorial pharmacogenomic guidance for psychiatric medications reduces overall pharmacy costs in a 1 year prospective evaluation. Curr Med Res Opin. 2015;31(9):1633-43. doi: 10.1185/03007995.2015.1063483. Epub 2015 Jul 23. PMID 26086890
- [Background] Hicks JK, Bishop JR, Sangkuhl K, Muller DJ, Ji Y, Leckband SG, Leeder JS, Graham RL, Chiulli DL, LLerena A, Skaar TC, Scott SA, Stingl JC, Klein TE, Caudle KE, Gaedigk A; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for CYP2D6 and CYP2C19 Genotypes and Dosing of Selective Serotonin Reuptake Inhibitors. Clin Pharmacol Ther. 2015 Aug;98(2):127-34. doi: 10.1002/cpt.147. Epub 2015 Jun 29. PMID 25974703